CLINICAL TRIAL: NCT02115633
Title: A Wearable "Balance Booster" - Stepping Closer to the Market
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RxFunction Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RxF-NIA-001; 2R44AG040865-02 (NIH)
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Distorted; Balance; Sensation Disorders; Peripheral Neuropathy; Neuropathy
MeSH Terms: conditions — Sensation Disorders; Peripheral Nervous System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Walkasins ON then OFF (Experimental): Subjects will first wear Walkasins and receive vibrotactile feedback that reflects real changes in center of pressure sway. Following a 1 hour rest period they will be retested with Walkasins turned off.
  Interventions: Device: Walkasins ON; Device: Walkasins OFF
- Walkasins OFF then ON (Experimental): Subjects will first wear Walkasins turned off and not receive any vibrotactile feedback. Following a 1 hour rest period they will be retested with Walkasins turned on.
  Interventions: Device: Walkasins ON; Device: Walkasins OFF

INTERVENTIONS:
Device: Walkasins ON — Subjects will be wearing a device that works as intended and provides real-time vibrotactile feedback that reflects center of pressure sway.
Device: Walkasins OFF — Subjects will be wearing a device that is turned off.

SUMMARY:
The overall goal of this project is to continue development and commercialization of a Wearable Sensory Prosthesis termed Walkasins. The device measures foot pressure through a thin sole insert, developed under National Institute on Aging (NIA) Small Business Innovation Research (SBIR) Phase I funding, and displays pressure information through a vibrotactile feedback array, placed around the lower leg, to help improve balance function. The device can replace lost foot pressure sensation in individuals with peripheral neuropathy who have balance problems.

DETAILED DESCRIPTION:
Our specific aims are to:

1. Revise and finalize design of Walkasins® based on accomplishments, user input, as well as reviewer criticism from our Phase 1 grant and manufacture 200 units of the device for clinical testing.

   Milestone 1: 200 units manufactured and ready for clinical testing under Aim 2. This goal is accomplished.
2. Investigate effects of using Walkasins on clinical outcomes related to gait, balance function and associated fall risk in a population of patients with sensory peripheral neuropathy and balance problems.

Hypotheses 1A-B: Patients who are trained to use Walkasins programmed to display relevant balance cues will attain higher gait speed and Functional Gait Assessment when compared to a matched cohort not using Walkasins.

Milestone 2: Data collection to assess clinical utility and safety of the Walkasins on patients briefly trained to use the device has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age diagnosed with Peripheral Neuropathy and who experience balance problems.
* Ability to perceive the Walkasins vibration feedback, understand and physically act on the vibration feedback.

Exclusion Criteria:

* Vibration to the skin is contraindicated by physician

  * Use of ankle foot orthotic that prevents attachment of Walkasins device
* Foot size smaller than Woman's 5 or larger than Men's 13

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-05; Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Koehler, PhD, Principal Investigator — Minneapolis VA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beninato M, Fernandes A, Plummer LS. Minimal clinically important difference of the functional gait assessment in older adults. Phys Ther. 2014 Nov;94(11):1594-603. doi: 10.2522/ptj.20130596. Epub 2014 Jun 19. PMID 24947198
- [Background] Hardy SE, Perera S, Roumani YF, Chandler JM, Studenski SA. Improvement in usual gait speed predicts better survival in older adults. J Am Geriatr Soc. 2007 Nov;55(11):1727-34. doi: 10.1111/j.1532-5415.2007.01413.x. Epub 2007 Oct 3. PMID 17916121
- [Background] Leddy AL, Crowner BE, Earhart GM. Functional gait assessment and balance evaluation system test: reliability, validity, sensitivity, and specificity for identifying individuals with Parkinson disease who fall. Phys Ther. 2011 Jan;91(1):102-13. doi: 10.2522/ptj.20100113. Epub 2010 Nov 11. PMID 21071506
- [Background] Lin JH, Hsu MJ, Hsu HW, Wu HC, Hsieh CL. Psychometric comparisons of 3 functional ambulation measures for patients with stroke. Stroke. 2010 Sep;41(9):2021-5. doi: 10.1161/STROKEAHA.110.589739. Epub 2010 Jul 29. PMID 20671244
- [Background] Perera S, Mody SH, Woodman RC, Studenski SA. Meaningful change and responsiveness in common physical performance measures in older adults. J Am Geriatr Soc. 2006 May;54(5):743-9. doi: 10.1111/j.1532-5415.2006.00701.x. PMID 16696738
- [Background] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Background] Wrisley DM, Kumar NA. Functional gait assessment: concurrent, discriminative, and predictive validity in community-dwelling older adults. Phys Ther. 2010 May;90(5):761-73. doi: 10.2522/ptj.20090069. Epub 2010 Apr 1. PMID 20360052
- [Background] Wrisley DM, Marchetti GF, Kuharsky DK, Whitney SL. Reliability, internal consistency, and validity of data obtained with the functional gait assessment. Phys Ther. 2004 Oct;84(10):906-18. PMID 15449976

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-one male community-dwelling veterans, ages 56-84, who experienced sensory peripheral neuropathy and balance problems, participated in the trial.
Groups:
- Walkasins On Then Off: Subjects will first wear Walkasins and receive vibrotactile feedback that reflects real changes in center of pressure sway. Following a 1-hour rest period they will be retested with Walkasins turned off.
  Walkasins On: Subjects will be wearing a device that works as intended and provides real-time vibrotactile feedback that reflects center of pressure sway.
  Walkasins Off: Subjects will be wearing a device that is turned off.
- Walkasins Off Then On: Subjects will first wear Walkasins turned off and not receive any vibrotactile feedback. Following a 1-hour rest period they will be retested with Walkasins turned on.
  Walkasins ON: Subjects will be wearing a device that works as intended and provides real-time vibrotactile feedback that reflects center of pressure sway.
  Walkasins OFF: Subjects will be wearing a device that is turned off.
Period: Overall Study
Arm/Group | Walkasins On Then Off | Walkasins Off Then On
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Walkasins On: Group A subjects first wore Walkasins and received real-time vibrotactile feedback that reflects real changes in center of pressure sway. Following a 1-hour rest period, they were retested with Walkasins turned off.
  The results for the Walkasins On state include all subjects, combining Group A, who were randomized to initially be tested with Walkasins turned on and then retested with walkasins turned off, and Group B, who were randomized to initially be tested with Walkasins turned off and then retested with Walkasins turned on.
- Walkasins Off: Group B subjects first wore Walkasins turned off and not receive any vibrotactile feedback. Following a 1-hour rest period, they were retested with Walkasins turned on.
  The results for the Walkasins Off state include all subjects, combining Group A, who were randomized to initially be tested with Walkasins turned on and then retested with walkasins turned off, and Group B, who were randomized to initially be tested with Walkasins turned off and then retested with Walkasins turned on.
- Total: Total of all reporting groups
Arm/Group | Walkasins On | Walkasins Off | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (7.1) | 71.6 (6.2) | 71.6 (6.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 16 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 31
Functional Gait Assessment (FGA) Score [Mean (Standard Deviation); unit: units on a scale] — The FGA is a reliable and valid measure of gait function related to postural stability and has been shown to be effective in classifying fall risk in older adults and predicting unexplained falls in community-dwelling older adults. The FGA includes a 10-item scale where each item is scored from 0 to 3 (3 = normal, 2 = mild impairment, 1 = moderate impairment, 0 = severe impairment). The maximum score is 30; the minimum score is 0. Higher scores represent a better outcome. An increase >4 is considered the MCID for community-dwelling elderly individuals (Beninato et al. 2014).
  units on a scale | 15.0 (4.5) | 15.4 (5.2) | 15.2 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Functional Gait Assessment (FGA)
Description: The Functional Gait Assessment (FGA) is a reliable and valid measure of gait function related to postural stability and has been shown to be effective in classifying fall risk in older adults and predicting unexplained falls in community-dwelling older adults (Wrisley, Marchetti et al. 2004; Wrisley and Kumar 2010). It has also been validated in stroke survivors (Lin, Hsu et al. 2010) and patients with Parkinson's disease (Leddy, Crowner et al. 2011) and has less flooring and ceiling effect than the Dynamic Gait Index (Lin, Hsu et al. 2010). The FGA includes a 10-item scale; each item is scored from 0 to 3 (3=normal, 2=mild impairment, 1=moderate impairment, 0=severe impairment). The maximum score is 30; minimum score, 0. Higher scores represent a better outcome. To be included in the count of participants, subjects' FGA scores needed to improve more than 4 points, which is the Minimally Clinically Important Difference (MCID) (Beninato et al. 2014).
Time Frame: During one test session < 3 hours
Measure: Count of Participants; unit: Participants
Groups:
- Walkasins OFF: Walkasins OFF: Subjects will wear Walkasins turned off and not receive any vibrotactile feedback.
Arm/Group | Walkasins ON | Walkasins OFF
Number analyzed (Participants) | 31 | 31
Participants | 17 | 7

2. Secondary Outcome: Four-Stage Balance Test >30s
Description: The 4-Stage Balance Test is part of the STEADI protocol recommended by the Centers for Disease Control and Prevention (CDC) to assess fall-risk in elderly individuals. It includes four gradually more challenging postures the subject performs; 1) Stand with feet side by side; 2) Stand with feet in semi-tandem stance; 3) Stand with feet in tandem stance; 4) Stand on one leg. Subjects pass if they can hold the stance for 10 seconds and then move on to the next stance. A fail during tasks 1, 2, or 3 indicates a high risk of falling, i.e., a total performance time of less than 30 seconds.
Time Frame: The assessment requires holding each stance for 10 seconds for a total of 40 seconds to pass.
Measure: Mean (Standard Deviation); unit: number of seconds stances held
Arm/Group | Walkasins ON | Walkasins OFF
Number analyzed (Participants) | 31 | 31
number of seconds stances held | 27.5 (7.4) | 25.6 (8.3)

3. Secondary Outcome: 10-Meter (10M) Walk Test (Measure of Gait Speed)--Number of Participants With Improvement to Normal Gait Speed
Description: The 10m-walk is routinely done in rehabilitation and has excellent reliability in chronic stroke patients. In addition, gait speed has been found to be an important predictor of survival in older adults (Hardy, Perera et al. 2006), further emphasizing its importance as a clinical outcomes measure. Gait speed (10-meter walk, timing only the middle 6 meters to allow for acceleration and deceleration) was assessed by instructing subjects to walk at their normal speed. A difference of 0.10m/sec is defined as the Minimally Clinical Important Difference (MCID) (Perera, Mody et al. 2006). Lower scores (# of seconds) on this measure indicate a better outcome. To be included in the count of participants, subjects' times on the 10M Walk Test needed to improve by more than 0.10m/sec, the MCID.
Time Frame: During one test session < 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Walkasins ON | Walkasins OFF
Number analyzed (Participants) | 31 | 31
Participants | 8 | 5

4. Secondary Outcome: Activities-Specific Balance Confidence Scale (ABC)
Description: Powell and Myers (1995) developed the Activities-specific Balance Confidence (ABC) Scale to detect levels of balance confidence in elderly persons. The ABC scale is a one-page questionnaire that asks questions about balance confidence when performing 16 different tasks. The items are rated on a scale of 0 to 100; a score of 0 indicates no confidence and a score of 100 indicates complete confidence when performing the task. The overall score is calculated by adding the individual items then dividing by the total number of items (16). The higher the score, the greater the person's balance confidence; thus, higher scores indicate that subjects are more confident of their balance. The ABC Scale was assessed only at baseline to document the level of balance confidence the subjects had before beginning the study intervention.
Time Frame: Measure was administered only at baseline during one test session <3 hours.
Measure: Mean (Standard Deviation); unit: score on a scale of 0-100
Groups:
- Walkasins ON Then OFF: Subjects will wear Walkasins and receive vibrotactile feedback that reflects real changes in center of pressure sway. Following a 1-hour rest period they will be retested with Walkasins turned off.
  Walkasins On: Subjects will be wearing a device that works as intended and provides real-time vibrotactile feedback that reflects center of pressure sway.
- Walkasins OFF: Subjects will first wear Walkasins turned off and not receive any vibrotactile feedback. Following a 1-hour rest period they will be retested with Walkasins turned on.
  Walkasins Off: Subjects will be wearing a device that is turned off.
Arm/Group | Walkasins ON Then OFF | Walkasins OFF
Number analyzed (Participants) | 15 | 16
score on a scale of 0-100 | 59.6 (19.3) | 64.7 (17.3)

ADVERSE EVENTS:
Time Frame: During a 3-hour testing period
Arm/Group | Walkasins ON Then OFF | Walkasins OFF Then ON
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16

LIMITATIONS AND CAVEATS:
Study limitations included the following:

* The study was not blinded.
* The study involved a small group consisting of males only.
* The study was only short-term (<3 hours).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT02115633/Prot_SAP_000.pdf